CLINICAL TRIAL: NCT05575648
Title: Investigation of Dual Task Performance in Children With Duchenne Muscular Dystrophy
Brief Title: Dual Task in Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Büşra Kayabınar, PhD candidate, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/13-45
Record Dates: First submitted 2022-10-08; First posted 2022-10-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Dual task; Balance; Gait
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duchenne Muscular Dystrophy (Other): Children who have been diagnosed with Duchenne Muscular Dystrophy.
  Interventions: Other: 10 meter walk test
- Healthy Subjects (Active Comparator): Children who have a normal motor and cognitive development.
  Interventions: Other: 10 meter walk test

INTERVENTIONS:
Other: 10 meter walk test — To assess the dual task performance of children 10 meter walk test will be used.

SUMMARY:
This study was planned to determine the effects of the dual-task performance of children with DMD with motor dysfunction and varying degrees of cognitive impairment compared to their healthy peers, to compare the dual-task performance of children with different functional levels, and to determine the relationship between parameters that may affect dual-task performance.

DETAILED DESCRIPTION:
Children who are at least 6 years old and who can walk 10 meters independently, whose Duchenne's muscular dystrophy (DMD) diagnosis has been confirmed as a result of genetic testing, will be included in the study. To determine dual-task performance, the 10-meter Walk Test will be performed with additional motor and cognitive tasks. Functional level (Brooke Lower Extremity Functional Classification), ambulation level (North Star Ambulation Rating), muscular performance and functions (6 Minute Walk Test), balance (Pediatric Berg Balance Scale and four square step test), fear of falling (Fear of Falling Questionnaire), gait (Gait in DMD Assessment Scale, Gait Quality and Independence Classification Scale in DMD, and Functional Evaluation Scale for Duchenne Muscular Dystrophy-Gait Domain (FES-DMD-GD)), cognitive level (Modified Mini-Mental State Test (MMDT)), independence and activity limitation (Pediatric Functional Independence Measure (WeeFIM) and ACTIVLIM), quality of life (The Pediatric Quality of Life Inventory (PedsQL)-Neuromuscular Module Turkish version PedsQL-3.0 Neuromuscular Module) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with DMD by a pediatric neurologist,
* Must be at least 6 years old and have the ability to walk 10 meters independently,
* Being able to cooperate with the instructions given by the physiotherapist,
* Not having undergone surgery in the last 6 months and not having any injuries,

Exclusion Criteria:

* Failure to cooperate with the physiotherapist who made the evaluations,
* Have had any injury and/or surgery in the last 6 months,
* Children without consent will not be included.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Dual task performance- 10 meter walk test | only baseline
  The time is measured after 10 meter walk completed
Dual task performance- 10 meter walk test with cognitive task | only baseline
  The time is measured after 10 meter walk with a cognitive (memory and mental) task completed
Dual task performance- 10 meter walk test with motor task | only baseline
  The time is measured after 10 meter walk with a motor task completed

SECONDARY OUTCOMES:
Functional level- Brooke Lower Extremity Functional Classification | only baseline
  It was developed using the classification method based on Vignos et al. to determine the functional status of the lower extremity. It consists of 10 different levels, ranging from Level 1 (walks independently and climbs stairs) to Level 10 (bound to bed).
Ambulation level- North star ambulatory assessment | only baseline
  It consists of an item that allows the evaluation of activities that children frequently use in their daily lives, such as "standing up from a chair", "climbing steps", "stepping down", "standing up", "running". Scoring; 2 = the activity is done unassisted, normally, 1 = the activity is done unassisted but in a modified form, and 0 = the activity cannot be done independently. The total score ranges from 0-34. A higher score indicates better ambulation and motor function. It is a practical and valid reliable scale for children with DMD.
Performance- 6 minutes walk test | only baseline
  The 6-minutes walk test (6 MWT), which is valid and reliable for DMD patients, will evaluate the walking function and physical capacity of children at the submaximal level. The distance the child walks for 6 minutes in a 25 m corridor will be recorded in meters. A physiotherapist will walk with the children during the test and track the time with a stopwatch. The 6 MWT is a simple test and considered an important outcome measure for children with DMD.
Balance - Pediatric berg balance scale | only baseline
  It is a test that functionally evaluates balance and consists of 14 parts, including parameters such as standing up from sitting, standing, transfers, taking steps, and turning. Each section is scored between 0-4 and the highest score that can be obtained from the scale is 56. High scores indicate good balance performance.
Balance - Four square step test | only baseline
  It is a valid and reliable test that has been used frequently in children in recent years to evaluate dynamic balance. Sticks, each 90 cm long, are placed on the floor to form 4 squares and the squares are numbered from 1 to 4. For the test to be completed successfully, the child must quickly move from one square to the next without touching the sticks. Performance is determined by measuring the test completion time in seconds. Shorter completion time means better dynamic balance.
Fear of falling - Pediatric Fear of Falling Questionnaire | only baseline
  Its validity and reliability have been established in children with DMD. The test consists of 34 items that question children's fear of falling during different activities in daily life. It is scored as "0=Never", "1=Sometimes", "2=Always" and the highest possible score is 68. Higher scores indicate greater fear of falling.
Fall frequency | only baseline
  How many times children have fallen in the last week (fall frequency) will be recorded.
Gait - Gait Evaluation Scale in Duchenne Muscular Dystrpohy | only baseline
  It consists of 10 items that examine the kinetic/kinematic condition of the foot, knee, hip, lumbar region, trunk, arm and head, support surface, walking speed and stride length, and each item is scored between 0 (worst) - 2 (best).
Gait - Gait Classification Scale in Duchenne Muscular Dystrpohy | only baseline
  It classifies gait with 5 levels, from Level 1 (Patient walks without compensation) to Level 5 (Patient cannot walk).
Gait - Functional Evaluation Scale for Duchenne Muscular Dystrophy-Gait Domain | only baseline
  It allows the compensatory movements of ambulatory children to be examined in detail through observation and provides a kinesiological analysis of gait by detecting and scoring compensatory movements. The scale consists of 3 parts: stance phase, swing phase and general compensatory movements. The points that can be obtained from the stance phase are between 0-23, the points that can be obtained from the swing phase are between 0-11, and the points that can be obtained from the general compensatory movements are between 0-13. Lower scores indicate good performance.
Cognitive level - Modified Mini Mental Test | only baseline
  The Mini Mental Test developed for adults was adapted to the pediatric population by making minor modifications. Test; It evaluates verbal responses including attention, orientation, memory and language skills, ability to obey verbal and written orders, write spontaneous sentences, and copy a complex drawing. The highest score that can be obtained from this test is 37, the lowest score is 0. The total score reaches a plateau at approximately 9-10 years of age and corresponds to the scores of healthy adults. Values below 27 points out of a total of 37 points in children over the age of 10 are indicative of mental retardation or dementia.
Activity of daily living - The Functional Independence Measure for Children (WeeFIM) | only baseline
  It consists of 6 sections and 18 items covering self-care, sphincter control, transfers, locomotion, communication, social and cognitive domains. Each item is scored between 7 (completely independent) and 1 (fully assisted) and the total score is determined as a minimum of 18 (fully dependent) and a maximum of 126 (completely independent).
Activity of daily living - ACTIVLIM | only baseline
  It is a scale developed to evaluate activity limitations in all neuromuscular diseases, including adult and childhood, and has Turkish validity and reliability. The scale includes 22 items that evaluate activities of daily living that require the use of the upper and lower extremities. Scoring; "0 = cannot do the activity", "1 = has difficulty in doing the activity", "2 = can do the activity easily" and according to this score, the patients are asked to describe their level of difficulty in performing each activity. The highest score that can be obtained from the test is 36, and higher scores indicate less activity limitations.
Quality of life - The Pediatric Quality of Life Inventory (PedsQL)-Neuromuscular Module Turkish version PedsQL-3.0 | only baseline
  This scale, which was found to be valid and reliable to evaluate the quality of life of children with neuromuscular disease, consists of 3 parts containing a total of 25 items. The first part contains 17 items about the disease, the second part contains 3 items about communication skills, and the third part contains 5 items about the family's financial resources and social support systems. The scale consists of a child personal report and a parent report for children aged 5-18, while only a parent report for children aged 2-4. Each item is scored between 4 (always a problem) - 0 (never a problem). Scoring is converted to 0=100, 1=75, 2=50, 3=25, 4=0. A higher score on the scale indicates a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Oznur YILMAZ, Prof, Study Director — Hacetteoe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No